CLINICAL TRIAL: NCT00816933
Title: Prospective Randomized Trial on the Assessment of Postoperative Outcomes According to the Number of Trocar During Laparoscopic Appendectomy
Brief Title: Trial on Postoperative Outcomes According to the Number of Trocar During Laparoscopic Appendectomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Wook Kim. MD, PhD, Professor & Chief
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HFHAPPE 01
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Appendicitis; Pain; Complications
Keywords: pain; operative times; complication; time to return for normal life; pain using VAS score
MeSH Terms: conditions — Appendicitis; Pain | interventions — Appendectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- one port (Experimental): Patients undergo one port appectomy. Skin incision about 2cm size is made upon umbilicus and dissection is performed to make opening. Then, wound retractcor(Alexis) is iserted on opening site and wound is extended. Rubber glove built-in three 5mm trocars is applied over wound retractor. Pneumoperitoneum is achieved via trocar and appendectomy is performed. After appendectomy, wound is repaired.
  Interventions: Procedure: appendectomy
- Three ports (Active Comparator): Paitents will undergo three port appendectomy. 10 mm trocar is inserted on umbilicus, and two 5mm trocas is inserted low abdomen, left flank respectively.
  Appendectomy is performed vis these trocas. After operation, wounds are repaired.
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Procedure: appendectomy — appendectomy according to the number of trocar

SUMMARY:
Appendicitis is the most common benign inflammatory disease that requires an operation.

Laparoscopic appendectomy using three trocar is generally performed, and reveals good surgical outcomes incluing less pain, early recovey, cosmetic effect et al. However, with using three trocar, there are some problems including pain around trocar insertion sites(three portions), wound infecton and scar at trocar insertion sites. For these reasons, more minimal invasive appendectomy is required, with development of laparoscopic instrument,eventually one port sppectomy is developed. So, the investigators assess post-operative Outcomes according to the Number of Trocar.

ELIGIBILITY:
Inclusion Criteria:

* Appendicitis (clinical or radilogical diagnosis)
* ASA < 4

Exclusion Criteria:

* Appendicitis with palpable mass( clinical or radilogical diagnosis)
* Patient has bleeding tendency
* Pregnant

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
post-operative pain | For 7days

SECONDARY OUTCOMES:
cosmetic effect | for 14days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, Holy Family Hospital, College of Medicine, The Catholic University of Korea, Bucheon-si, Gyunggi Do, South Korea

REFERENCES:
- [Derived] Kye BH, Lee J, Kim W, Kim D, Lee D. Comparative study between single-incision and three-port laparoscopic appendectomy: a prospective randomized trial. J Laparoendosc Adv Surg Tech A. 2013 May;23(5):431-6. doi: 10.1089/lap.2012.0284. Epub 2013 Mar 8. PMID 23473061
- [Derived] Lee J, Baek J, Kim W. Laparoscopic transumbilical single-port appendectomy: initial experience and comparison with three-port appendectomy. Surg Laparosc Endosc Percutan Tech. 2010 Apr;20(2):100-3. doi: 10.1097/SLE.0b013e3181d84922. PMID 20393336